CLINICAL TRIAL: NCT02382744
Title: A Comparison of Ultrasound-Guided and Ultrasound-Guided With Nerve Stimulation Saphenous Nerve Blockade Utilizing the Transsartorial Approach
Brief Title: Saphenous Nerve Block for Foot and Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Scott Bell, Dr. Scott Bell, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H14-02912
Record Dates: First submitted 2015-02-18; First posted 2015-03-09 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-09

CONDITIONS: Saphenous Nerve Block
Keywords: Saphenous Nerve; Nerve Block; Ultrasound guided; Neurostimulation; Regional Anesthesia; Ropivacaine; Foot Surgery; Nerve Stimulation; Ankle Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Guidance (Experimental): Saphenous nerve block placed using ultrasound guidance alone
  Interventions: Device: Ultrasound Guidance
- Ultrasound Guidance + nerve stimulation (Experimental): Saphenous nerve block placed using ultrasound guidance and nerve stimulation
  Interventions: Device: Ultrasound guidance + nerve stimulation

INTERVENTIONS:
Device: Ultrasound Guidance — Ultrasound guidance will be used to place a saphenous nerve block
  Arms: Ultrasound Guidance
Device: Ultrasound guidance + nerve stimulation — Ultrasound guidance and nerve stimulation will be used to place a saphenous nerve block
  Arms: Ultrasound Guidance + nerve stimulation

SUMMARY:
Patients undergoing foot and ankle surgery have the option of having a nerve block administered by their Anesthesiologist. The nerve block numbs the foot and results in less post-operative nausea and vomiting, and better pain control. Two different techniques for blocking the saphenous nerve to the foot have been described and are both commonly used at St. Paul's hospital. The goal of this study is to compare the success rates of these two techniques.

DETAILED DESCRIPTION:
Purpose / Hypothesis This clinical study is a prospective, controlled, randomized, single-blinded trial designed to investigate the hypothesis that ultrasound-guided blockade of the saphenous nerve in conjunction with nerve stimulation has a higher success rate when compared to ultrasound alone. These research interventions represent what is considered to be an improvement on the standard practice at St. Paul's, which is to block the saphenous nerve with one of any number of saphenous nerve blocks, using a number of different techniques (i.e. ultrasound-guided, nerve stimulation, blind field block); the effectiveness of which has been inconsistent. The purpose of this study is to identify if one technique has a great success rate over another, which would ultimately result in increased success rates of saphenous nerve blocks and patient care.

Study Design The study will be a randomized, single-blinded trial of 80 subjects who are undergoing foot and ankle surgery. Informed consent will be obtained from all study subjects. Subjects will be randomized to one of two saphenous nerve block techniques to be administered by an experienced regional anesthesiologist at St. Paul's Hospital. Once the nerve block is completed the success will be evaluated by an investigator blinded to the procedure. Once the 30min evaluation is completed anesthetic care will be provided according to regular institutional practice and at the discretion of the attending anesthesiologist. The subject will then be contacted at 2 and 7 days after block administration to assess for delayed complications.

Intravenous access will be gained and non-invasive blood pressure measurements will be recorded every five minutes. Continuous electrocardiography and oxygen saturation monitoring will be maintained throughout the procedure and for at least 60 minutes afterwards. Light sedation will be provided, with the goal of maintaining verbal contact with the subject throughout the procedure. Where clinically appropriate, the study block may be preceded by an ultrasound-guided popliteal sciatic nerve block at the discretion of the attending anesthesiologist.

Saphenous nerve blockade will be preformed using a transsartorial approach. Subjects in both groups will be positioned prone. The ultrasound probe will be placed in the transverse plane on the medial aspect of the thigh 3-5cm cephalad to the superior border of the patella (area marked). An attempt will then be made to identify the saphenous nerve, which runs deep to the sartorius muscle within the subsartorial fascial plane. The nerve will appear hyperechoic, round or oval shaped. The anesthesiologist will have a maximum scan time of 3 minutes prior to needle entry. Up to 5 mL of 1% Lidocaine will be used for skin infiltration of the injection site. The block will then be preformed as to the protocols below depending on group allocation. A thirty minute evaluation of the saphenous nerve block will occur during the normal monitoring period after the placement of a block.

Following completion of the thirty-minute evaluation, anesthetic care will be provided according to regular institutional practice and at the discretion of the attending anesthesiologist. This may include spinal or general anesthesia.

All subjects will be contacted by telephone at two and seven days post procedure for a follow up interview to assess for delayed complications associated with the procedure.

The medications used for the nerve blocks in the study will include only ropivacaine 0.5% and lidocaine 1%. For subject sedation, midazolam and fentanyl will be used. None of these medications are considered study drugs; rather they are commonly used anesthetic medications. While used in the study, these drugs themselves are not being investigated. The same medications will be used on subjects not enrolled in the study.

Study Treatment Group 1 - Saphenous nerve block using ultrasound guidance The needle will be placed with the needle tip in close proximity (1-2 mm) of the target structures (the saphenous nerve if visible or in the subsartorial facial plane of the sartorius muscle if the nerve is not visible). A total of 10 mL of 0.5% ropivacaine will be used for the block. Before injection of any local anesthetic a gentle aspiration will be preformed, with a second aspiration after 5 mL of ropivacaine has been injected. Once injection of local anesthetic has commenced small needle adjustments are allowed to enhance spread. This will be done at the discretion of the regional anesthesiologist performing the block.

Study Treatment Group 2 - Saphenous nerve blockade using ultrasound guidance and nerve stimulation The needle will be place with the needle tip in close proximity (1-2 mm) of the target structure (the saphenous nerve if visible or in the subsartorial fascial plane if the nerve is not visible). The Pajunk MultiStim SENSOR nerve stimulator will then be turned on, starting at 1.0 milliamp (mA) until a tapping sensation is elicited in the medial or anterior aspect of the ankle. The amplitude of the nerve stimulator will then be gradually decreased with maintenance of the tapping sensation by making small adjustments in needle location. The end-point for nerve localization will be a tapping sensation in the area of the medial malleolus at ≤ 0.6 mA. The anesthesiologist will have a maximum search time of 5 minutes from needle entry to elicitation of the tapping sensation. Once a tapping sensation is elicited in the ≤ 0.6 mA range, 10 mL of 0.5% ropivacaine will be injected at the site. If a tapping sensation is elicited but not ≤ 0.6 mA within 5 minutes then 10 mL of 0.5% ropivacaine will be injected at the site where the lowest amplitude tapping sensation was elicited. If no tapping sensation is elicited from the subject after 5 minutes, an injection of 10 mL of ropivacaine will be made below the Sartorius muscle in the subsartorial fascial plane. Before injection of any local anesthetic a gentle aspiration will be preformed, with a second aspiration after 5 mL of ropivacaine has been injected. Once injection of local anesthetic has commenced small needle adjustments are allowed to enhance spread. This will be done at the discretion of the regional anesthesiologist performing the block.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing foot and ankle surgery
2. Aged 19-80
3. Normal sensation in saphenous nerve distribution in both legs
4. Provided written informed consent.
5. Body Mass Index <38 kg/m2

Exclusion Criteria:

1. Subject refusal
2. A known history of allergy, sensitivity or any other form of reaction to local anesthetics of amide type
3. Suspected inability to comply with study procedures, including language difficulties or medical history and/or concomitant disease (i.e. skin infection as the site of needle insertion), as judged by the investigator. Reason for exclusion will be recorded.
4. A neurological and/or vascular condition, which may preclude eligibility for peripheral nerve blockade (i.e. peripheral neuropathy) as judged by the investigator. Reason for exclusion will be recorded.
5. Subjects on therapeutic anticoagulation or coagulopathy at the time of nerve blockade.
6. Previous inclusion in this study.
7. Participation in other clinical studies during this study or in the 14 days prior to admission to this study.
8. Surgeon refusal (e.g. the surgeon does not want a nerve block for the subject). Reason for exclusion will be recorded.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bell, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsui BC, Ozelsel T. Ultrasound-guided transsartorial perifemoral artery approach for saphenous nerve block. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):177-8; author reply 178. doi: 10.1097/AAP.0b013e31819a273e. No abstract available. PMID 19282716
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Lopez AM, Sala-Blanch X, Magaldi M, Poggio D, Asuncion J, Franco CD. Ultrasound-guided ankle block for forefoot surgery: the contribution of the saphenous nerve. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):554-7. doi: 10.1097/AAP.0b013e3182611483. PMID 22854395
- [Background] Chen J, Lesser J, Hadzic A, Resta-Flarer F. The importance of the proximal saphenous nerve block for foot and ankle surgery. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):372. doi: 10.1097/AAP.0b013e318295596a. No abstract available. PMID 23788076
- [Background] Head SJ, Leung RC, Hackman GP, Seib R, Rondi K, Schwarz SK. Ultrasound-guided saphenous nerve block--within versus distal to the adductor canal: a proof-of-principle randomized trial. Can J Anaesth. 2015 Jan;62(1):37-44. doi: 10.1007/s12630-014-0255-1. Epub 2014 Oct 22. PMID 25337966
- [Background] Benzon HT, Sharma S, Calimaran A. Comparison of the different approaches to saphenous nerve block. Anesthesiology. 2005 Mar;102(3):633-8. doi: 10.1097/00000542-200503000-00023. PMID 15731603
- [Background] Chi J, Greensmith JE. Saphenous nerve block technique with neurostimulation. Reg Anesth Pain Med. 2007 Nov-Dec;32(6):548-9. doi: 10.1016/j.rapm.2007.08.007. No abstract available. PMID 18035315
- [Background] Comfort VK, Lang SA, Yip RW. Saphenous nerve anaesthesia--a nerve stimulator technique. Can J Anaesth. 1996 Aug;43(8):852-7. doi: 10.1007/BF03013038. PMID 8840065
- [Background] van der Wal M, Lang SA, Yip RW. Transsartorial approach for saphenous nerve block. Can J Anaesth. 1993 Jun;40(6):542-6. doi: 10.1007/BF03009739. PMID 8403121
- [Derived] Montgomery SH, Shamji CM, Yi GS, Yarnold CH, Head SJ, Bell SC, Schwarz SK. Effect of Nerve Stimulation Use on the Success Rate of Ultrasound-Guided Subsartorial Saphenous Nerve Block: A Randomized Controlled Trial. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):25-31. doi: 10.1097/AAP.0000000000000522. PMID 27902645

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasound Guidance and Nerve Stimulation: Saphenous nerve block placed using ultrasound guidance and nerve stimulation
  Ultrasound guidance and nerve stimulation: Ultrasound guidance and nerve stimulation will be used to place a saphenous nerve block
Period: Overall Study
Arm/Group | Ultrasound Guidance | Ultrasound Guidance and Nerve Stimulation
Started | 40 | 40
Allocated | 40 | 40
Analyzed | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guidance | Ultrasound Guidance and Nerve Stimulation | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15) | 53 (14) | 52 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 18 | 11 | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26 (3) | 25 (4) | 25 (4)
American Society of Anesthesiologists (ASA) physical status [Number; unit: participants] — ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: A moribund patient who is not expected to survive without the operation
  (For reference, see https://www.asahq.org/resources/clinical-information/asa-physical-status-classification-system)
  participants
    I or II | 37 | 33 | 70
    III to V | 3 | 7 | 10
Type of surgery [Number; unit: participants]
  Foot/ankle joint reconstruction/fusion/arthrodesis | 15 | 24 | 39
  Arthroscopy/debridement | 7 | 7 | 14
  Mass/hardware removal | 9 | 3 | 12
  Fracture fixation | 5 | 3 | 8
  Tendon repair/transfer | 4 | 2 | 6
  Amputation | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Block Success
Description: Complete absence of sensation to pinprick at two different anatomic areas of the saphenous nerve at thirty minutes
Time Frame: 30 minutes post nerve block
Measure: Number; unit: participants
Groups:
- Ultrasound Guidance + Nerve Stimulation: Saphenous nerve block placed using ultrasound guidance and nerve stimulation
  Ultrasound guidance and nerve stimulation: Ultrasound guidance and nerve stimulation will be used to place a saphenous nerve block
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants | 18 | 22
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; We sought to detect an increase in the rate of complete absence of sensation to pinprick 30 min following ultrasound-guided subsartorial saphenous nerve blockade to 90% from an assumed baseline of 64% as extrapolated from our previous study (cf. Head SJ et al. 2015) at β = 0.2. The required minimum sample size at α = 0.05 (one-sided) was 30 patients in each group. To be conservative, we aimed to enroll a total of 80 patients; Test type: Superiority or Other; p = 0.25, Fisher Exact — One-sided P-value based on the lack of plausibility that additional nerve stimulation would worsen sensory blockade rates; Difference between proportions (%) = 10.0, 95% CI 2-sided [-11.9 to 31.9]

2. Secondary Outcome: Block Failure Rate
Description: Persistent sensation in the saphenous nerve distribution at 30 minutes (i.e., absence of any evidence of blockade [decreased or complete absence of sensation] at both areas: normal sensation.
Time Frame: 30 minutes post nerve block
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  Normal sensation | 1 | 3
  Decreased or no sensation | 39 | 37
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; This contingency-table type analysis (Fisher Exact test) compares the two groups, "Ultrasound Guidance" and "Ultrasound Guidance and Nerve Stimulation", as far as the two categorical outcomes are concerned, "block failure at 30 minutes post nerve block" versus "no block failure at 30 minutes post nerve block"; Test type: Superiority or Other; p = 0.62, Fisher Exact — Two-sided P-value

3. Secondary Outcome: Any Evidence of Blockade (Decreased or Complete Absence of Sensation)
Description: Participants with any evidence of blockade (decreased or complete absence of sensation) at the two different anatomic areas in the distribution of the saphenous nerve (2 cm proximal to the medial malleolus and 10 cm distal to the medial tibial condyle)
Time Frame: 30 min
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants | 39 | 37
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; Test type: Superiority or Other; p = 0.62, Fisher Exact

4. Secondary Outcome: Incomplete Block Rate
Description: incomplete [decreased only] loss of sensation in the saphenous nerve distribution at 30 minutes at both areas of assessment
Time Frame: 30 minutes post nerve block
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  Decreased sensation | 21 | 15
  Normal or no sensation | 19 | 25
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; This contingency-table type analysis (Fisher Exact test) compares the two groups, "Ultrasound Guidance" and "Ultrasound Guidance and Nerve Stimulation", as far as the two categorical outcomes are concerned, "incomplete block at 30 minutes post nerve block" versus "no incomplete block at 30 minutes post nerve block"; Test type: Superiority or Other; p = 0.26, Fisher Exact — Two-sided P-value

5. Secondary Outcome: Speed of Onset for Nerve Block (Complete Blockade)
Description: Median (Kaplan-Meier curve "survival") time required to reach complete absence of sensation to pinprick at the two different anatomic areas of assessment in the distribution of the saphenous nerve (2 cm proximal to the medial malleolus and 10 cm distal to the medial condyle of the tibia).
Time Frame: 30 minutes post nerve block
Population: Participants with complete absence of sensation to pinprick at the two different anatomic areas of assessment in the distribution of the saphenous nerve (2 cm proximal to the medial malleolus and 10 cm distal to the medial condyle of the tibia)
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 18 | 22
Minutes | 25.0 [20.0 to 30.0] | 17.5 [15.0 to 25.0]
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; To assess speed of onset, sensation to pinprick in the distribution of the saphenous nerve was assessed for each patient every 5 min until complete sensory loss was noted, or until 30 min had elapsed. To compare the two groups in speed of onset on the basis of these data, we constructed Kaplan-Meyer "survival" curves for the times to onset of sensory blockade and compared the underlying time-to-event data with the log-rank test; Test type: Superiority or Other; p = 0.12, Log Rank; "Median survival" ratio = 0.70, 95% CI 2-sided [0.38 to 1.31] — Numerator, group "Ultrasound Guidance"; denominator, group, "Ultrasound Guidance + Nerve Stimulation"

6. Secondary Outcome: Rate of Success of Elicitation of a Tapping Sensation
Description: successful elicitation of any "tapping" sensation in the saphenous nerve distribution within the 5 min stimulation time limit
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40
participants | 32

7. Secondary Outcome: Mean Minimum Stimulation Current
Description: the mean minimum stimulation current magnitude to elicit "tapping" sensation in the saphenous nerve distribution (cf. 3.2.3 below)
Time Frame: 5 minutes
Population: Participants in the "Ultrasound Guidance and nerve stimulation" group with available data
Measure: Mean (95% Confidence Interval); unit: mA
Arm/Group | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 26
mA | 0.39 [0.31 to 0.48]

8. Secondary Outcome: Rate of Success of Elicitation of a Tapping Sensation at < 0.6 Milliampere (mA)
Description: Successful elicitation of "tapping" sensation in the saphenous nerve distribution at ≤ 0.6 mA
Time Frame: 5 minutes
Population: Participants in the "Ultrasound Guidance and nerve stimulation" group with successful stimulation and available current magnitude data
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance and Nerve Stimulation
Number analyzed (Participants) | 26
participants | 25

9. Secondary Outcome: Time Required to Administer Block
Description: The time required for the block to be completed (from scanning to removal of needle)
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
s | 207 (76) | 314 (125)
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Difference between means (s) = 107, 95% CI 2-sided [61 to 153]

10. Secondary Outcome: Immediate Complications
Description: Any complications as a result of block placement (e.g. local anesthetic toxicity, hematoma, pain etc.)
Time Frame: 60 minutes post block completion
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  Local anesthetic systemic toxicity | 0 | 0
  Hematoma | 0 | 0
  Pain on needle manipulation | 1 | 0
  Paresthesia | 3 | 2
  Positive aspiration (of blood) | 0 | 1
  Pruritus of the blocked leg in saph. n. distrib. | 1 | 0
  Transient increase in pain in medial malleolus | 1 | 0

11. Secondary Outcome: Delayed Complications
Description: Any complication as a results of nerve block placement (e.g. persistent paresthesia, nerve injury)
Time Frame: 7 days post operative
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  Paresthesia | 0 | 1
  Other | 0 | 0

12. Post Hoc Outcome: Speed of Onset for Any Blockade in the Area 2 cm Proximal to the Medial Malleolus Only
Description: Median (Kaplan-Meier curve "survival") time required to reach any evidence of sensory blockade (decreased or complete absence of sensation) in the area 2 cm proximal to the medial malleolus only
Time Frame: 30 min
Population: Participants with any evidence of sensory blockade (decreased or complete absence of sensation) in the area 2 cm proximal to the medial malleolus only
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 35 | 36
Minutes | 30.0 [20.0 to 30.0] | 17.5 [15.0 to 25.0]
Statistical Analysis 1: Comparison: Ultrasound Guidance vs Ultrasound Guidance + Nerve Stimulation; Test type: Superiority or Other; p = 0.02, Log Rank; "Median survival" ratio = 0.58, 95% CI 2-sided [0.37 to 0.93] — Numerator, group "Ultrasound Guidance"; denominator, group, "Ultrasound Guidance + Nerve Stimulation"

13. Post Hoc Outcome: Sensory Blockade Scores by Individual Assessment Area: Medial Malleolus
Description: Sensation to pinprick with an 18 gauge blunt needle was assessed individually at the two different anatomic areas in the distribution of the saphenous nerve: Here, the results are reported for the area 2 cm proximal to the medial malleolus only
Time Frame: 30 min
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  2 = absent sensation | 24 | 31
  1 = decreased sensation | 14 | 5
  0 = normal sensation (no block) | 2 | 4

14. Post Hoc Outcome: Sensory Blockade Scores by Individual Assessment Area: Medial Tibial Condyle
Description: Sensation to pinprick with an 18 gauge blunt needle was assessed individually at the two different anatomic areas in the distribution of the saphenous nerve: Here, the results are reported for the area 10 cm distal to the medial tibial condyle only
Time Frame: 30 min
Measure: Number; unit: participants
Arm/Group | Ultrasound Guidance | Ultrasound Guidance + Nerve Stimulation
Number analyzed (Participants) | 40 | 40
participants
  2 = absent sensation | 21 | 23
  1 = decreased sensation | 17 | 14
  0 = normal sensation (no block) | 2 | 3

15. Post Hoc Outcome: Response Versus Lack of Response to Nerve Stimulation and Block Failure Rate
Description: Percentage of block failure (persistent sensation in the saphenous nerve distribution at 30 minutes -- i.e., absence of any evidence of blockade [decreased or complete absence of sensation] at both areas: normal sensation) among participants in the Ultrasound Guidance and Nerve Stimulation group with response versus no response to nerve stimulation
Time Frame: 30 min
Measure: Number; unit: participants
Groups:
- Responders to Nerve Stimulation: Participants in the Ultrasound Guidance and Nerve Stimulation group with response to nerve stimulation
- Non-responders to Nerve Stimulation: participants in the Ultrasound Guidance and Nerve Stimulation group with no response to nerve stimulation
Arm/Group | Responders to Nerve Stimulation | Non-responders to Nerve Stimulation
Number analyzed (Participants) | 32 | 8
participants
  Block failure (normal sensation) | 0 | 3
  No block failure (decreased or no sensation) | 32 | 5
Statistical Analysis 1: Comparison: Responders to Nerve Stimulation vs Non-responders to Nerve Stimulation; This contingency-table type analysis (Fisher Exact test) compares the two arms, "Patients with response to nerve stimulation" and "Patients with lack response to nerve stimulation", as far as the two categorical outcomes are concerned, "block failure at 30 minutes post nerve block" versus "no block failure at 30 minutes post nerve block"; Test type: Superiority or Other; p = 0.0057, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data were collected immediately (i.e., on the day of the intervention/postoperative day 0); on postoperative days 2 and 7, patients were contacted via telephone to enquire about the presence of any delayed complications. In case of presence of any delayed complications at the day 7 follow-up, patients were to be contacted every 7 days until symptom resolution, and further investigations and/or management were to be provided at this time.
Description: As noted above, all patients were systematically followed up via telephone to enquire about the presence of any delayed complications/adverse events.
Arm/Group | Ultrasound Guidance | Ultrasound Guidance and Nerve Stimulation
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 3/40 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Guidance (N=40) | Ultrasound Guidance and Nerve Stimulation (N=40)
Paresthesia (on regional nerve block needle manpulation/advancement) (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) — Common localized event during regional anesthesia (traditionally deliberately sought for nerve localization); transient and reversible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No